CLINICAL TRIAL: NCT04751513
Title: Auricular Acupressure Improves Oxaliplatin-induced Peripheral Neuropathy and Quality of Life
Brief Title: Auricular Acupressure : Improves Oxaliplatin-induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001339B0
Record Dates: First submitted 2021-01-25; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Oxaliplatin-induced Peripheral Neuropathy; Chemotherapy
Keywords: colorectal cancer; chemotherapy; Oxaliplatin-induced peripheral neuropathy; auricular acupressure; pain; quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: This study will conduct a randomized controlled trial by randomly assigning all participants to either the experimental group receiving auricular acupressure and usual care or the control group only receiving usual care. This study provides an auricular acupressure for eight weeks, and assesses the immediate and carry-over effects. These assessments happen biweekly during the intervention period, two weeks after the intervention period, as well as one month after the end of the chemotherapy course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive acupressure on six auricular points.
  Interventions: Other: auricular acupressure
- Control group (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Other: auricular acupressure — Pressure on auricular point of Shenmen (TF4), Sympathesis (AH6a), Subcortex (AT4), Endocrine (CO18), finger (SF1), and toe (AH2) of the ear.
  Arms: Experimental group

SUMMARY:
Oxaliplatin-induced peripheral neuropathy (OIPN) is a common adverse effect that becomes worse as the drug dose accumulation impacts cancer patients' daily activities and quality of life.The result of this study will determine the immediate effects of the 8-week auricular acupuncture intervention on alleviating the participants' OIPN symptoms and enhancing their quality of life. This study will continue to evaluate the carry-over effects of auricular acupuncture after the chemotherapy course ends.

DETAILED DESCRIPTION:
Objectives:

Oxaliplatin-induced peripheral neuropathy (OIPN) is a common adverse effect that becomes worse as the drug dose accumulation impacts cancer patients' daily activities and quality of life. This study aims to evaluate the immediate and carry-over effects of auricular acupressure on OIPN symptoms and quality of life for colorectal cancer patients.

Methods :

This randomized trial will recruit 76 participants with colorectal cancer and OIPN from the oncology outpatient department in Taiwan. The control group will receive usual care, whereas the experimental group will receive usual care in addition to auricular acupressure for 8 weeks. Outcomes will be assessed by using the chemotherapy-induced peripheral neuropathy assessment tool, neuropathic pain symptom inventory, pain visual analogue scale, and the European Organization for research and treatment of cancer-quality of life questionnaire-core 30. These assessment tools are used before the intervention, biweekly during the intervention, 2 weeks after the intervention, and one month after the end of the chemotherapy course.

Hypothesis:

Ultimately, the result of this study will determine the immediate effects of the 8-week auricular acupuncture intervention on alleviating the participants' OIPN symptoms and enhancing their quality of life. This study will continue to evaluate the carry-over effects of auricular acupuncture after the chemotherapy course ends.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients who are above the age of 20 years
* Have experiencing Oxaliplatin induced peripheral neuropathy
* Must be able to communicate
* Willing to fill out the inform consent

Exclusion Criteria:

* Symptoms of peripheral neuropathy caused by diabetes mellitus
* Symptoms of peripheral neuropathy caused by genetic disease
* Symptoms of peripheral neuropathy caused by spinal cord injury
* Symptoms of peripheral neuropathy caused by alcoholism
* With wounds on ears
* Allergy to latex (the tapes for the auricular acupressure include latex)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
National Cancer Institute Common Terminology Criteria for Adverse Events v5.0[NCI-CTCAE v5.0] | This assessment tool is used at baseline, change from baseline after 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and one month followed by completing the chemotherapy course.
  For the severity of peripheral neuropathy symptoms caused by Oxaliplatin chemotherapy.
Chemotherapy-induced Peripheral Neuropathy Assessment Tool(CIPNAT) | This assessment tool is used at baseline, change from baseline after 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and one month followed by completing the chemotherapy course.
  This questionnaire is a self-assessment of the patient. It is divided into four parts: 1. The severity of symptoms; 2. The degree of trouble the symptom causes; 3. The frequency of symptoms; 4. The symptom's degree of interference in daily life.
Neuropathic Pain Symptom inventory (NPSI) | This assessment tool is used at baseline, change from baseline after 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and one month followed by completing the chemotherapy course.
  This questionnaire mainly used to assess the symptoms and severity of neuropathic pain. This questionnaire consists of four parts: 1. spontaneous and persistent pain, 2. spontaneous paroxysmal pain, and 3. Induced pain and paresthesia
Visual Analogue Scale (VAS) | This assessment tool is used at baseline, change from baseline after 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and one month followed by completing the chemotherapy course.
  This study uses the Visual Analogue Scale (VAS) for pain. The patient will Self-assess the pain intensity based on their subjective feelings and current pain state.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30 version 3.0 (EORTC QLO-C30). | This assessment tool is used at baseline, change from baseline after 8 weeks, 10 weeks, and one month followed by completing the chemotherapy course.
  The purpose of this questionnaire is to evaluate the impact of the overall quality of life of cancer patients after suffering from cancer or receiving treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan